CLINICAL TRIAL: NCT01927172
Title: AirSonea Wheeze Detection Study - Multipart Clinical Performance Assessment to Determine Agreement on Wheeze Detection Between AirSonea™ Versus Physician Auscultation and an Expert Panel.
Brief Title: AirSonea Wheeze Detection Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: iSonea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: iS-2013-Wz
Record Dates: First submitted 2013-08-02; First posted 2013-08-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- AirSonea (Other): Use of AirSonea to detect wheeze sounds.
  Interventions: Device: AirSonea

INTERVENTIONS:
Device: AirSonea
  Other Names: No intervention, AirSonea is an adjuct to physician/clinician auscultation.

SUMMARY:
The purpose of this study is to determine if the AirSonea device provides an objective assessment of breath sounds for the presence of wheeze in both medical and home environments.

ELIGIBILITY:
Inclusion Criteria:

* Part I: Participants presenting to an Acute Care Setting with an exacerbation of asthma or chronic obstructive pulmonary disease symptoms
* Part II: Volunteer participants without asthma
* Part III: Participants with asthma
* For all parts of study

  * Age: 18 years or older
  * Participant has signed an Informed Consent after having the Study explained to them.

Exclusion Criteria:

* Any medical finding by the physician that would exclude the patient from participating.
* < than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Device Efficacy | 1 day
  Device wheeze detection as compared to physician wheeze detection via auscultation.

SECONDARY OUTCOMES:
Wheeze Rate break points | Up to 1 week
  Wheeze Rate break points for the user of rescue inhalers